CLINICAL TRIAL: NCT02788617
Title: A Prospective, Non-interventional, Multicenter, Clinical Study to Evaluate the Efficacy of the Diafert G-CSF ELISA as an Adjunct to Morphological Assessment in Predicting Embryos' Potential to Develop to the Blastocyst Stage
Brief Title: Evaluation of the Efficacy of Diafert in Predicting Embryos' Potential to Develop to the Blastocyst Stage
Status: Completed | Type: Observational
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: DFT-MD-05
Record Dates: First submitted 2016-04-26; First posted 2016-06-02 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human follicular fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non treatment group: This is a non-interventional study in which embryo selection is performed according to standard of care. The Diafert output, the granulocyte colony-stimulating factor (G-CSF) concentration in follicular fluid (FF), will be recorded but will not be used in patient management, ie, values will not be used for embryo selection in the assisted reproduction procedure.
  Interventions: Device: Diafert

INTERVENTIONS:
Device: Diafert — The Diafert output, the G-CSF concentration in FF, will be recorded but will not be used in patient management.

SUMMARY:
This prospective study will evaluate the efficacy of Diafert as an adjunct to morphological assessment in predicting embryos' potential to develop to the blastocyst stage on Day 5.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before initiation of any study procedures
* Be a female outpatient, ≥ 18 years of age at the time of informed consent
* Have at minimum 10 mature egg follicles as of the last transvaginal ultrasound following hormonal stimulation
* Eligible to allow embryos to develop through day 5 before implantation or freezing

Exclusion Criteria:

* Presence of ovarian endometriotic cyst
* Presence or history of diagnosed severe endometriosis (i.e. stage IV the revised American Fertility Society classification for endometriosis).
* Need for pre-implantation genetic diagnosis/screening of embryos
* Use of time-lapse embryo imaging
* Employee or immediate relative of an employee of Forest Research Institute, Inc., any of its affiliates or partners, or the study center

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female outpatients involved in an assisted reproduction procedure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Number of Embryos that achieve the blastocyst stage of development at Day 5 as determined by morphological assessment using the SART criteria | Day 5
  The status of each embryo will be assessed by an independent panel of 5 embryologists through visual inspection using the Society for Assisted Reproductive Technology (SART) criteria to determine if each embryo has achieved the blastocyst stage of development or not.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Somers, PhD, Study Director — Allergan
Locations (9):
- United States (9):
  - Huntington Reproductive Center, Encino, California
  - Women's Medical Research Group, Clearwater, Florida
  - InVia Fertility Specialists, Hoffman Estates, Illinois
  - Institute for Reproductive Health, Cincinnati, Ohio
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Dallas - Fort Worth Fertility Associates, Dallas, Texas
  - Houston Fertility Institute, Houston, Texas
  - Utah Fertiity Center, Pleasant Grove, Utah
  - Reproductive Care Center, Sandy City, Utah